CLINICAL TRIAL: NCT00253032
Title: PRIMA Study: Pain Relief Investigation of NeuroModulation Therapy in an Adult Population: A Double Blind, Randomized, Multicenter, Placebo Controlled Trial.
Brief Title: Pain Relief Investigation of NeuroModulation Therapy in Adult Humans
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Fralex Therapeutics (Industry)
Collaborators: PharmaNet (Industry)
Other Study IDs: F05001
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2006-03-03 (Estimated); Status verified 2006-03

CONDITIONS: Chronic Musculoskeletal Pain

INTERVENTIONS:
Device: PRIMA

SUMMARY:
The study is being performed to determine the efficacy and safety of Fralex Neuromodulation Therapy (F-NMT), delivered by the Fralex PRIMA device, in reducing chronic musculoskeletal pain.

Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Derived] Sepulveda-Sanchez JM, Gil-Gil M, Alonso-Garcia M, Vaz Salgado MA, Vicente E, Mesia Barroso C, Rodriguez Sanchez A, Duran G, De Las Penas R, Munoz-Langa J, Velasco G, Hernandez-Lain A, Hilario A, Navarro Martin M, Benavides M, Oleaga L, Cantero Montenegro D, Ruano Y, Sanchez-Gomez P, Martin-Soberon MC, Morales-Llombart R, Pachon V, Pineda E. Phase II Trial of Palbociclib in Recurrent Retinoblastoma-Positive Anaplastic Oligodendroglioma: A Study from the Spanish Group for Research in Neuro-Oncology (GEINO). Target Oncol. 2020 Oct;15(5):613-622. doi: 10.1007/s11523-020-00754-6. PMID 33025213